CLINICAL TRIAL: NCT07264283
Title: The Progressive Supranuclear Palsy Clinical Trial Platform - Regimen B: LM11A-31
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Adam Boxer (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Alzheimer's Therapeutic Research Institute (Other); University of Southern California (Other); Massachusetts General Hospital (Other); University of California, San Diego (Other); Alzheimer's Clinical Trials Consortium (Other); PharmatrophiX Inc. (Industry)
Responsible Party: Sponsor-Investigator, Adam Boxer, Endowed Professor in Memory and Aging, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATRI-015-B; R01AG085029 (NIH)
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: PSP - Progressive Supranuclear Palsy
Keywords: PSP; Placebo-Controlled; Double-Blind; Regimen Specific Appendix; LM11A-31; Tau Protein; Oral treatment; Disease modifying; P75 neurotrophin receptor; Synaptic resilience
MeSH Terms: conditions — Supranuclear Palsy, Progressive; Frontotemporal Dementia | interventions — LM11A-31

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Regimen B: LM11A-31 (Experimental)
  Interventions: Drug: LM11A-31
- Matching Placebo (Placebo Comparator)
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: LM11A-31 — LM11A-31 is administered orally twice daily.
  Arms: Regimen B: LM11A-31
Drug: Matching Placebo — Matching placebo is administered orally twice daily.
  Arms: Matching Placebo

SUMMARY:
The Progressive Supranuclear Palsy Clinical Trial Platform (PTP) is a multi-center, multi-regimen clinical trial evaluating the safety and efficacy of investigational products for the treatment of PSP. Regimen B will evaluate the safety and efficacy of a single study drug, LM11A-31, in participants with PSP.

DETAILED DESCRIPTION:
The Progressive Supranuclear Palsy Clinical Trial Platform (PTP) is designed as a perpetual platform trial. This means that there is a single Master Protocol dictating the conduct of the trial. The PTP Master Protocol is registered as NCT07173803. Once a participant enrolls into the Master Protocol and meets all eligibility criteria, the participant will be eligible to be randomized into any currently enrolling regimen. All participants will have an equal chance to be randomized to all regimens that are active at the time of screening. If a participant is randomized to Regimen B: LM11A-31, participants will complete a baseline assessment and be randomized in a 3:1 ratio to either active LM11A-31 or matching placebo. Participants must first enroll into the Master Protocol and be eligible to participate in the Master Protocol before being able to be randomly assigned to Regimen B. For a list of enrolling sites, please see the PTP Master Protocol under NCT07173803.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of possible or probable PSP Richardson's Syndrome as defined by the 2017 Movement Disorder Society (MDS) criteria.
2. Presence of PSP symptoms for ≤5 years at screening (based on the best judgment of the site PI).
3. Mini-Mental State Examination (MMSE) score at screening of ≥25.
4. Able to walk at least 10 steps with minimal assistance (e.g., one arm for safety, but not postural support).
5. Stable doses of permitted medications as described per protocol for 30 days prior to screening.
6. Resides at home or in the community (assisted living is acceptable).
7. As assessed by the site PI, participant is likely to be able to comply with the protocol for the duration of the study, and has adequate vision, hearing (hearing aid permitted), and literacy (English or Spanish) sufficient for compliance with the required testing procedures.

Exclusion Criteria:

1. Females who are breastfeeding or pregnant (as documented by a urine pregnancy test) during screening, or plan to become pregnant during the study.
2. Females of childbearing potential who did not use a highly effective method of contraception within 28 days of screening and/or are not willing to use a highly effective method of contraception for the duration of their participation in the study.
3. Lacks good venous access such that multiple blood draws would be precluded.
4. Weighs less than 40kg, or more than 136kg at screening.
5. Blood transfusion within 4 weeks of screening.
6. Contraindications to MRI studies, including metal (ferromagnetic) implants, a cardiac pacemaker that is not compatible with MRI, and/or severe claustrophobia.
7. Screening MRI scan showing structural evidence of alternative pathology not consistent with PSP that could explain a substantial portion of the participant's symptoms as indicated by the central MRI read.
8. Any unstable and/or clinically significant medical condition likely to hamper the evaluation of safety and/or efficacy of study drug (e.g., clinically significant reduction in serum B12 or folate levels, clinically significant abnormalities of thyroid function, stroke, or other cerebrovascular or cardiovascular conditions), as per the site PI's judgment.
9. History of severe allergic reaction (e.g., anaphylaxis) including but not limited to: severe allergic reaction to previous vaccines, foods, and/or medications.
10. Hospitalization within 30 days prior to screening or baseline.
11. Infections or major surgical procedures within 3 months prior to screening, judged to be clinically significant by the site PI.
12. Myocardial infarction within 1 year prior to baseline, unstable angina pectoris, symptomatic congestive heart failure.
13. History of cancer within the past 5 years other than treated skin squamous cell carcinoma, basal cell carcinoma, and melanoma in-situ, localized prostate cancer not requiring treatment, or prostate or breast cancer, which have been fully removed and are considered cured.
14. History or presence of immunological or inflammatory conditions, including neurological disorders, meningitis or meningoencephalitis.
15. History or presence of epilepsy requiring ongoing use of antiepileptic medications. Antiepileptic medications are permitted for pain or psychiatric use per the protocol.
16. DSM-5 criteria for drug or alcohol abuse or dependence currently met within the past 5 years.
17. Clinically significant abnormal vital signs including sustained sitting blood pressure >160/100 mm Hg.
18. Diabetes mellitus with hemoglobin A1c (HbA1c) levels of ≥8.0%.
19. Known history of human immunodeficiency virus (HIV-1 or 2).
20. Known history of acute/chronic hepatitis B or C unless treated curatively.

Ages: 41 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2029-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Disease progression | 52 weeks
  Change in disease severity as measured by the 15-item modified Progressive Supranuclear Palsy Rating Scale (mPSPRS-15) in which the minimum score is 0 and the maximum score is 52, with higher scores indicating a worse outcome.

SECONDARY OUTCOMES:
Disease progression | 52 weeks
  Change in disease severity as measured by the 10-item modified Progressive Supranuclear Palsy Rating Scale (mPSPRS-10) in which the minimum score is 0 and the maximum score is 30, with higher scores indicating a worse outcome.
Disease progression | 52 weeks
  Change in disease severity as measured by the 28-item Progressive Supranuclear Palsy Rating Scale (28-item PSPRS) in which the minimum score is 0 and the maximum score is 100, with higher scores indicating a worse outcome.
Experiences of daily living | 52 weeks
  Change in experiences of daily living over time as measured by the Cortical Basal ganglia Functional Scale (CBFS) in which the minimum score is 0 and the maximum score is 124, with higher scores indicating a worse outcome.
Activities of daily living | 52 weeks
  Change in activities of daily living over time as measured by the Schwab and England Activities of Daily Living Scale (SE-ADL) in which the minimum score is 0% and the maximum score is 100%, with lower scores indicating a worse outcome.
Disease severity | 52 weeks
  Change in disease severity over time as measured by the Clinical Global Impression of disease severity (CGIds) using a 7-point scale, ranging from 1 (normal, not ill) to 7 (extremely ill), with a higher score indicating a worse outcome.
Disease progression | 52 weeks
  Change in disease severity over time as measured by the Clinical Global Impression of Change (CGIC) using a 7-point scale, ranging from 1 (very much improved) to 7 (very much worse), with a score of 4 indicating no change.
Health-related quality of life | 52 weeks
  Change in quality of life over time as measured by the EuroQoL 5 Dimension - 5 Level (EQ-5D-5L) questionnaire in which the minimum score is 0 and the maximum score is 1, with lower scores indicating a worse outcome.
Brain volume | 52 weeks
  Change in volume in midbrain, pontine and other regions over time as measured by volumetric MRI.
Neurodegeneration | 52 weeks
  Change in plasma neurofilament light chain (NfL) concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Boxer, MD, PhD, Principal Investigator — University of California, San Francisco; Irene Litvan, MD, Principal Investigator — University of California, San Diego; Julio Rojas-Martinez, MD, PhD, Principal Investigator — University of California, San Francisco; Anne-Marie Wills, MD, Principal Investigator — Massachusetts General Hospital

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol